CLINICAL TRIAL: NCT00944372
Title: An Open-Label, Multi-Center, Phase 4 Study to Evaluate the Effect of Age (Geriatric) and Renal Function on the Safety, Efficacy (Sensitivity, Specificity) and Pharmacokinetics of OctreoScan in Patients Referred for Scintigraphy of All Solid Tumors With a High Suspicion of Containing Somatostatin Receptor Positive Tissue
Brief Title: Study to Evaluate the Effect of Age (Geriatric) and Kidney Function on the Safety, Efficacy and Pharmacokinetics of OctreoScan in Patients Who Have New or Recurrent Tumors
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment was difficult
Sponsor: Mallinckrodt (Industry)
Responsible Party: James Brodack, Ph.D., Mallinckrodt
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 0050-02-763
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Solid Tumors
Keywords: Tumor; somatostatin receptor
MeSH Terms: conditions — Neoplasms | interventions — pentetreotide; Indium-111

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Group 1 (Experimental): Control, age greater than or equal to 18 with normal renal function
  Interventions: Drug: Indium In-111 pentetreotide
- Group 2 (Experimental): Age 18 to less than 65 with mild renal impairment
  Interventions: Drug: Indium In-111 pentetreotide
- Group 3 (Experimental): Age 18 to less than 65 with moderate to severe renal impairment
  Interventions: Drug: Indium In-111 pentetreotide
- Group 4 (Experimental): Age 18 to less than 65 with end stage renal impairment
  Interventions: Drug: Indium In-111 pentetreotide
- Group 5 (Experimental): Age 65 to less than 75 with mild renal impairment
  Interventions: Drug: Indium In-111 pentetreotide
- Group 6 (Experimental): Age 65 to less than 75 with moderate to severe renal impairment
  Interventions: Drug: Indium In-111 pentetreotide
- Group 7 (Experimental): Age 65 to less than 75 with end stage renal impairment
  Interventions: Drug: Indium In-111 pentetreotide
- Group 8 (Experimental): Age greater than or equal to 75 with mild renal impairment
  Interventions: Drug: Indium In-111 pentetreotide
- Group 9 (Experimental): Age greater than or equal to 75 with moderate to severe renal impairment
  Interventions: Drug: Indium In-111 pentetreotide
- Group 10 (Experimental): Age greater than or equal to 75 with end stage renal impairment
  Interventions: Drug: Indium In-111 pentetreotide

INTERVENTIONS:
Drug: Indium In-111 pentetreotide — Single intravenous injection of 222MBq (6.0 mCi) Indium In-111 pentetreotide
  Other Names: OctreoScan; In-111

SUMMARY:
The objective of this study was to evaluate the effect of age (geriatric) and renal function on the safety, efficacy and pharmacokinetics of OctreoScan at the recommended clinical dose in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 18 years of age and older.
2. If female and of childbearing potential, patients must have a negative pregnancy test within 24 hours of study drug administration. In addition, all female patients of childbearing potential must agree to use a medically accepted method of contraception throughout the study.
3. If deemed necessary by the Principal Investigator, patients entering the pharmacokinetic population must be willing to be housed within the investigational facility for a minimum of 24 hours following drug administration.
4. Patients (when able) or legally authorized representatives must have the ability to understand the requirements of the study and provide written consent to participate and agree to abide by the study requirements.
5. Patients must have tumor localization by conventional imaging methods prior to enrollment (i.e., CT, MRI, US, angiogram).
6. Patients referred for scintigraphy of solid tumors with a high suspicion of containing somatostatin receptor positive tissue.
7. Patients with first-time tumors must be scheduled for a tissue biopsy. A tissue sample will be sent to the core laboratory for conventional histology and immunohistochemistry analysis.
8. Patients with recurrent tumors or progressive tumors must have previous biopsy results documented, with previous biopsy tissue obtainable for immunohistochemistry analysis.

Exclusion Criteria:

1. Patients receiving Sandostatin LAR < 21 days prior to dosing or Sandostatin Immediate Release (IM) < 24 hours prior to dosing.
2. Patients who have received any investigational drug within 30 days of admission into this study or plan to participate in a clinical study prior to the end of this study's monitoring period (patients on a research protocol using an approved drug are accepted).
3. Patients who are pregnant, breastfeeding or lactating.
4. Patients with a medical condition, serious intercurrent illness, or extenuating circumstance that would significantly decrease study compliance, including all prescribed follow-up.
5. Patients scheduled to undergo any scintigraphy within 7 days prior to study participation or PET scanning within 24 hours prior to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-07; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Assessment of OctreoScan diagnostic sensitivity for detecting tumor(s) confirmed as somatostatin receptor positive by biopsy with immunohistochemistry analysis | Through 24 hours post dose

SECONDARY OUTCOMES:
Assessment of OctreoScan diagnostic sensitivity for detecting tumor(s) confirmed as somatostatin receptor positive using previously biopsied tissue for immunohistochemistry analysis | Through 24 hours post dose

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Miami, Jackson Memorial Hospital, Miami, Florida
  - University of Iowa Medical Center, Iowa City, Iowa
  - Louisiana State University, Division of Hem/Onc, New Orleans, Louisiana
  - Hospital of University of Pennsylvania, Division of Nuclear Medicine, Philadelphia, Pennsylvania